CLINICAL TRIAL: NCT06580145
Title: Leucine as a Probe of Kynurenine-Induced Glutamate and Neural Circuit Dysfunction in Midlife Depression
Brief Title: Leucine in Midlife Depression
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ebrahim Haroon, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00006751; R01MH132059 (NIH)
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Major Depression
Keywords: Major Depression; Kynurenine (KYN) pathway; Leucine in Midlife Depression; inflammation
MeSH Terms: conditions — Depressive Disorder, Major; Inflammation | interventions — Leucine; Lysine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-leucine (Experimental)
  Interventions: Drug: L-leucine
- L-lysine (Active Comparator)
  Interventions: Drug: L-lysine

INTERVENTIONS:
Drug: L-leucine — L-leucine is an essential amino acid used to competitively inhibit kynurenine uptake into the brain via the large neutral amino acid transporter (LAT1).
  The proposed dose for L-leucine is 4.31 g/day, administered orally.
  Other Names: Leucine
  Arms: L-leucine
Drug: L-lysine — L-lysine monohydrochloride is also an essential amino acid. It serves as an active comparator to control for general effects on brain protein synthesis and enters the brain through separate cationic amino acid transporters.
  The proposed dose for L-lysine is 6 g/day, administered orally
  Other Names: Lysine
  Arms: L-lysine

SUMMARY:
The study aims to investigate the effects of a 6-week leucine challenge on brain chemistry, connectivity, and behavior in people with midlife depression.

The researchers will compare the leucine and an active comparator arm (lysine) for 6 weeks.

DETAILED DESCRIPTION:
Major depression is a common and serious mental health condition that can severely impact a person's quality of life. Some symptoms, like loss of pleasure in activities and slowed movements, may be signs that the depression will be harder to treat. These symptoms are also linked to a higher risk of dementia later in life.

Scientists think that long-term, low-level inflammation in the body may contribute to depression, especially in middle-aged adults. This inflammation may affect areas of the brain involved in feeling good and controlling movement.

One way inflammation might lead to depression is through a process in the body called the kynurenine pathway. When activated by inflammation, this pathway can produce substances that are toxic to brain cells. These toxins can disrupt how brain cells communicate and function.

Leucine, a nutrient found in some foods, may help block these toxic substances from entering the brain. While animal studies have shown promise, we do yet know if leucine can help humans with depression.

To find out, researchers are planning a 6-week study in middle-aged adults with depression and signs of inflammation. Half the participants will take leucine supplements, while the other half will take a different supplement (lysine) for comparison. The study will use brain scans and symptom assessments to see if leucine improves brain function and reduces depression.

If successful, this research could point to new ways to treat depression, especially in cases that do not respond well to current treatments. It may also help reduce the risk of dementia in people with depression. This study is an important step in understanding how inflammation affects mental health and in developing new treatments to help people feel better.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent
* Diagnosis of major depression per Structured Interview for DSM-V (SCID-V)
* Moderate to severe depression- Inventory of Depressive Symptoms - Self Reported (IDS-SR score >34).
* SHAPS score >30 on the 0-56 scale
* Body mass index (BMI) between 20-35 kg/m2
* Plasma CRP >1 mg/L
* No contraindications to MRI
* Availability of friends or family for transportation after lumbar puncture procedure
* Clinically significant findings on EKG
* Patient Health Questionnaire (PHQ-9) score greater than 10
* Willingness to adopt contraceptive measures. Persons exempt from contraception requirements are:

  * Persons assigned male at birth
  * Persons assigned female at birth who:

    * have undergone a hysterectomy or bilateral oophorectomy; or
    * have been naturally postmenopausal for at least 24 consecutive months (i.e., has NOT had menses at any time in the preceding 24 consecutive months)

Exclusion Criteria:

* Leucine-Specific:

  * History of maple syrup urine disease
  * Risk of hypoglycemia (unstable diabetes)
  * History of vitamin B6 deficiency, relative
* Lysine-Specific:

  * On calcium supplements, relative
  * History of renal/gall stones (could cleared by a primary care provider)
* Cognitive:

  --Cognitive impairment (MMSE score <28)
* Psychiatric Disorders:

  * Lifetime diagnosis of psychotic disorders.
  * Current mania/hypomania.
  * Substance use disorder in the last 6 months.
  * Active suicidal ideation:
  * Psychiatric hospitalization in the past year.
  * Suicide attempts within the last five years.
  * Scores >3 on the Columbia Suicide Severity Rating Scale (C-SSRS)
  * Binge eating in the absence of mood symptoms increases.
  * Primary diagnosis of severe DSM-V79 anxiety disorders.
  * Primary diagnosis of DSM-V PTSD (if severity exceeds major depression).
  * Primary diagnosis of DSM-V obsessive-compulsive disorders.
  * Significant personality disorders with multiple hospitalizations or suicide attempts.
  * Developmental disorders (e.g., ADHD).
* Concomitant medications:

  * Immune-active medications (e.g., non-steroidal anti-inflammatory agents).
  * Antibiotics and immunizations in the past 2 weeks.
  * Topical or inhaled steroids within the past week.
  * Oral/parenteral steroids in the last 6 months.
  * Supplements that impact the immune system (e.g., omega-3, probiotics) within the past 2 weeks.
  * Psychotropic medications within the last 4 weeks (8 weeks for fluoxetine).
  * Daily use of sedative-hypnotics, benzodiazepines, and opiates.
* Medical Disorders:

  * Unstable medical disorders (frequent provider or medication changes).
  * Lifetime diagnosis/treatment of cancers (excluding basal cell carcinoma).
  * Lifetime diagnosis/treatment of autoimmune disorders.
  * Lifetime exposure to chemotherapeutic agents.
* MRI Considerations:

  -- Location and quantity of metallic objects safe to MR
* Concomitant Treatment for Depression:

  -- Treatments with antidepressant medications or those with antidepressant effects (dopamine supplements).
* Treatment for General Medical Conditions (GMCs):

  * Stabilized medications are allowed if maintained at the same dose during the trial.
  * Multiple recent changes in concomitant medications reviewed by the study PI
* Population

  * Pregnant women.
  * Children.
  * Prisoners.
  * Individuals unable to consent

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Change in Glutamate | Baseline, Week 1, Week 6
  Change in glutamate measured by magnetic resonance spectroscopy (MRS) in the basal ganglia in the leucine challenged group compared with the lysine-challenged group.

SECONDARY OUTCOMES:
Change in blood oxygen level dependent (BOLD) oscillatory coherence | Baseline, Week 1, Week 6
  Changes in blood oxygen level dependent (BOLD) oscillatory coherence, measured by regional homogeneity (ReHo) in the basal ganglia and its functional connectivity to the dorsomedial prefrontal cortex (dmPFC) between the two groups.
Changes in effort discontinuation ability | Baseline, Week 1, Week 6
  The Effort Expenditure for Rewards Task (EEfRT) will be utilized measure to assess motivational deficits related to anhedonia. The EEfRT is a computerized task where participants choose between easy (low-effort, low-reward) and hard (high-effort, high-reward) tasks, with varying probabilities of reward receipt.
  An increase in the proportion of high-effort choices over time would indicate improved motivation and potentially increased willingness to expend effort to achieve rewards
Change in anhedonia | Baseline, Week 1, Week 6
  The Snaith-Hamilton Pleasure Scale - Clinician Version (SHAPS-C) will be administered by trained clinicians at baseline and specified follow-up visits as outlined in the Schedule of Assessments. The SHAPS-C is a 14-item scale measuring consummatory (enjoyment) aspects of anhedonia.
  Lower scores indicate a greater capacity for pleasure, while higher scores reflect more severe anhedonia. An alternate version of SHAPS (SHAPS) is available as a self-rated version, where participants will rate themselves on a scale. The self-ratings are added to generate a total score, which has similar characteristics as those for SHAPS-C.
Change in MRS myo-inositol | Baseline, Week 1, Week 6
  Change in MRS myo-inositol (mI) in the basal ganglia 6 between the leucine and lysine groups will be assessed.
Changes in psychomotor slowing | Baseline, Week 1, Week 6
  Psychomotor slowing will be assessed as a tertiary outcome using neurocognitive tests. These include the Finger Tapping Task (FTT), Simple and Choice Reaction Time tasks from the Cambridge Automated Neuropsychological Test Assessment Battery (CANTAB), Digit Symbol Substitution Test (DSST), and Trail Making Tests A and B. The FTT measures pure motor function, while the Reaction Time tasks on CANTAB assess the speed and accuracy of responses. The DSST evaluates information processing speed, and the Trail Making Tests assess cognitive flexibility and task-switching abilities. Improved performance on these tasks, indicated by faster completion times and increased accuracy, would suggest a reduction in psychomotor slowing.

CONTACTS AND LOCATIONS:
Overall Officials: Ebrahim Haroon, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
PI will share individual de-identified participant data, including data dictionaries according to institutional, state, and Federal regulations. This aligns with Emory University's commitment to transparency and compliance with NIH guidelines, which support making research data widely available while ensuring participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be available starting at publication and remain accessible for a period specified in our Data Management and Sharing Plan (DMSP), as required by NIH, institutional, and state regulations. This typically means the data will be available for several years post-publication to facilitate ongoing research.
Access Criteria: Data will be shared with qualified researchers who submit an approved research proposal. PI requires that the researchers sign a Data Transfer Agreement (DTA) to ensure compliance with ethical and legal standards.
  The team will use a secure data repository (NIH DataArchive) to share the data, as specified in our DMSP. This ensures that data is accessible while maintaining security and compliance with Emory's and NIH's data-sharing policies
URL: https://nda.nih.gov/